CLINICAL TRIAL: NCT03002987
Title: Active Pregnancy Policy at Work. Greater Wellbeing and Lower Sickness Absence
Acronym: AGp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Luise Mølenberg Begtrup, MD, phD, postdoc, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AGp2016
Record Dates: First submitted 2016-12-19; First posted 2016-12-26 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Pregnancy; Sickness Absence; Occupational Exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention, education (Active Comparator): Education of leaders (3 hours) in how to implement Active Pregnancy policy at their departements/workplaces
  Interventions: Behavioral: Active Pregnancy policy
- control (No Intervention): as usual

INTERVENTIONS:
Behavioral: Active Pregnancy policy — Education (3 hours) of leaders in how to implement Active pregnancy policy at their departments/work places
  Arms: Intervention, education

SUMMARY:
In a cluster randomized design it will be investigated whether teaching local leaders how to implement active pregnancy policy results in less sickness absence among their pregnant employees. Further it will be investigated to what extent Active pregnancy policy is implemented at the departments and whether it results in higher sense of security and wellbeing among the pregnant employee. Finally the cost and benefits of the intervention will be analyzed.

DETAILED DESCRIPTION:
Background: The majority of Danish women work during their reproductive years. Sickness absence among pregnant women is frequent; more than one third of Danish women are on longterm sick leave during pregnancy. Sick leave has been found associated with occupational exposures and studies have shown that adjustment in exposure can reduce sick leave in pregnancy indicating that there are potential preventive initiatives.

Design and outcomes: In a cluster randomized design it will be investigated whether teaching local leaders how to implement active pregnancy policy results in less sickness absence among their pregnant employees. It will further be investigated to what extent Active pregnancy policy is implemented at the departments and whether it results in higher sense of security and wellbeing among the pregnant employee. Finally the cost and benefits of the intervention will be analyzed.

The study takes place at hospitals in the two regions on Zealand, Denmark (The Capital region of Denmark and Region Zealand) and in the daycare sector in 2 municipalities located in The Capital region of Denmark. The randomization will be at the level of departments, which will be randomized to either intervention or control:

Intervention: The leaders are invited to a 3 hours seminar, where they will be taught in how to implement active pregnancy policy at their department.

Control: as usual

All employees at the involved departments getting pregnant during the year of intervention will be included in the study. They are to answer a questionnaire at 28th week of gestation and their days of sick leave during pregnancy will be recorded. All leaders at the departments are to answer two questionnaires, one before randomization and one after intervention.

The intervention: At the 3 hours seminar the leaders will receive education containing: 1) Updates on evidence on pregnancy and risk of occupational exposures, 2) information about the rules in the area and the leader's responsibilities, 3) Answers and solutions to frequent issues relating pregnant employees at work and 4) Introduction to Active Pregnancy policy.

The content of Active Pregnancy Policy: A congratulation letter to the pregnant employee inviting her to a meeting. At the meeting her job task will be discussed and fears and worries taken hand on. The aim is to adjust the job tasks to the employee and her special need during her pregnancy. During the pregnancy the leader regularly evaluate with the pregnant employee on how it goes and if there are needs for other or further adjustments. A minimum of 3 planned meetings have to be held during the pregnancy. Further the leader shall inform the other employees at the workplace about the arrangements made with the pregnant employee.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy during intervention period, employed at one of the included departments/workplaces

Exclusion Criteria:

* not being able to understand, write and read Danish

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 866 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
pregnancy related sick leave | one year (intervention period)
  difference in pregnancy related sick leave between the two randomized groups. In days and the proportion of pregnant employee with longterm sick leave (> 4 weeks)

SECONDARY OUTCOMES:
To what extent Active pregnancy policy is implemented at the departments/workplaces | one year (intervention period)
  Difference between the two randomized groups in relation to the proportion of pregnant employees who experienced active pregnancy policy (different parts: Received congratulation letter, had scheduled meetings discussing the possible occupational exposures, adjustment of work tasks)
Wether active pregnancy policy lead to higher sense of security and wellbeing among the pregnant employees | one year
  Difference between the two randomized groups in relation to the experience of security and wellbeing among the pregnant employees. Using the WHO-5 and variables concerning the psychosocial work environment
cost effectiveness of the intervention | one year
  calculating the costs of the intervention: 1)Holding the seminars (place, salary for teachers, food supply etc.) 2) time used (the leaders salary) attending the seminars, 3) Teaching material and the cost of resources used at the departments (control vs. intervention): 1) time used hiring temporary employees, 2) time used talking with pregnant employees, 3) time used changing the work tasks of the pregnant employee, 4) Salary to hired temporary employees.

CONTACTS AND LOCATIONS:
Overall Officials: Luise Moelenberg Begtrup, MD, Principal Investigator — Department of occupational Medicine, Bipspebjerg Hospital
Locations (1):
- Department of occupational and evironmental medicine, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Begtrup LM, Malmros P, Brauer C, Soegaard Toettenborg S, Flachs EM, Hammer PEC, Bonde JP. Manager-oriented intervention to reduce absence among pregnant employees in the healthcare and daycare sector: a cluster randomised trial. Occup Environ Med. 2021 Jan 12:oemed-2020-106794. doi: 10.1136/oemed-2020-106794. Online ahead of print. PMID 33436380